CLINICAL TRIAL: NCT03470649
Title: Effect of Intravenous Iron Isomaltoside on Postoperative Anemia in Patients Underwent Total Knee Arthroplasty: A Single-blind Randomized Controlled Trial
Brief Title: Effect of IV Iron Isomaltoside on Postoperative Anemia in Total Knee Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-1709-079-885
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Anemia; Knee Arthropathy
MeSH Terms: conditions — Anemia | interventions — iron isomaltoside 1000; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patients in this group would receive Iron Isomaltoside 1000 (Monofer®) after main procedure of total knee arthroplasty. The dose of iron isomaltoside would be determined based on the patient's body weight.
  Interventions: Drug: Iron Isomaltoside 1000
- Control (No Intervention): Patients in this group would receive 100ml of normal saline after main procedure of total knee arthroplasty.

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Iron Isomaltoside 1000 would be intravenously administrated to treatment group after main procedure of total knee arthroplasty.
  Other Names: treatment
  Arms: Treatment

SUMMARY:
Postoperative anemia is a frequent complication after total knee arthroplasty, with an incidence of 87%. Iron supplementation is known to be effective in treatment and prevention of postoperative anemia. The investigators examined the effect of intravenous iron isomaltoside (Monofer®) administration on postoperative anemia and transfusion requirements in patients undergoing total knee arthroplasty.

Participants undergoing total knee arthroplasty will be randomly assigned to treatment group or control group. After main procedure of total knee arthroplasty, iron isomaltoside 1000 (Monofer®) or normal saline will be intravenously administered depending on the group assigned. The dose of iron isomaltoside will be determined based on patient's body weight using the manufacturer's recommendation. Serum hemoglobin, hematocrit, iron, ferritin, transferrin saturation, and phosphorus level will be checked at preoperative day, postoperative day 1, 7, and 30.

The primary outcome is the incidence of postoperative anemia at 30 days after surgery. Secondary outcomes included the incidence and amount of red blood cell transfusion during admission period, hospital length of stay, the incidence of surgical site infection, and quality of life during postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing total knee arthroplasty

Exclusion Criteria:

* bilateral total knee arthroplasty
* hematochromatosis or hemosiderosis
* hemolytic anemia
* history of drug allergy
* liver cirrhosis or hepatitis
* systematic lupus erythematosus
* rheumatic arthritis
* allergic disease
* history of transfusion within one month from surgery
* parturient

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Postoperative anemia | 30 days after surgery
  Incidence of postoperative anemia at 30 days after surgery

SECONDARY OUTCOMES:
Transfusion | During admission period for surgery, an average of 2 weeks
  Incidence and amount of red blood cell transfusion during admission
Hemoglobin | 1 day, 7 days, and 30 days after surgery
  serum hemoglobin level (g/dL)
Hematocrit | 1 day, 7 days, and 30 days after surgery
  Hematocrit level (%)
Iron | 1 day, 7 days, and 30 days after surgery
  serum iron level (μg/dL)
Ferritin | 1 day, 7 days, and 30 days after surgery
  serum ferritin level (ng/mL)
Transferrin saturation | 1 day, 7 days, and 30 days after surgery
  Transferrin saturation (%)
Phosphorus | 1 day, 7 days, and 30 days after surgery
  Serum phosphorus level (mg/dL)
Surgical site infection | During admission period for surgery, an average of 2 weeks
  Incidence of surgical site infection
Hospital length of stay | During admission period for surgery, an average of 2 weeks
  Hospital length of stay (days)
Quality of life using EQ-5D | 30 days after surgery
  Assessment of quality of life during postoperative periods using EQ-5D (EuroQol-5 Dimension) questionaire
Quality of life using FACT-An | 30 days after surgery
  Assessment of quality of life during postoperative periods using FACT-An (The Functional Assessment of Cancer Therapy-Anemia) questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Pf., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yoo S, Bae J, Ro DH, Han HS, Lee MC, Park SK, Lim YJ, Bahk JH, Kim JT. Efficacy of intra-operative administration of iron isomaltoside for preventing postoperative anaemia after total knee arthroplasty: A randomised controlled trial. Eur J Anaesthesiol. 2021 Apr 1;38(4):358-365. doi: 10.1097/EJA.0000000000001389. PMID 33259451